CLINICAL TRIAL: NCT01013883
Title: Long Term Outcomes in Patients With Heart Failure
Brief Title: The Darlington Retrospective Outpatient Study
Acronym: DROPSY
Status: Completed | Type: Observational
Sponsor: County Durham and Darlington NHS Foundation Trust (Other Government)
Collaborators: University of Durham (Other)
Responsible Party: Principal Investigator, Rajender Singh, Research registrar, County Durham and Darlington NHS Foundation Trust
Other Study IDs: RajPh.D2066
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure
Keywords: systolic dysfunction; diastolic dysfunction; mortality; treatment; heart rate
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- systolic dysfunction: patients having left ventricular systolic dysfunction on echocardiography
- distolic heart failure: patients with clinical heart failure and preserved LV systolic dysfunction

SUMMARY:
Having heart failure means the heart is unable to pump blood around the body effectively. This reduces life expectancy and hinders normal daily activities. Heart failure affects about one million people in the UK; it is a major cause of death but it is often undetected and under-treated. If diagnosed and treated properly, the symptoms of heart failure can be well controlled and the length and quality of life can be improved.

Two drugs (called ACE-inhibitors and beta-blockers) help patients to live longer and suffer fewer consequences of heart failure. These drugs should be offered to all patients although this does not happen consistently for a variety of reasons. Doctors specialising in heart failure may help patients make better informed decisions about treatments and other aspects of care.

The purpose of this research is to explore the diagnosis, management and outcome of patients with heart failure who are referred to the one stop diagnostic heart failure clinic between Jan 2002 and Dec 2007. This study will provide vital information about diagnosis, initiation and titration of evidence based medication in the hospital, their follow in the primary care and subsequent patient outcome in terms of mortality.

DETAILED DESCRIPTION:
Case notes of all the patients who were referred to the one stop diagnostic heart failure clinic during the period (Jan 2002- Dec 2007) will be reviewed and subjects who were found to have signs and symptoms of the Heart failure will be identified.

This cohort of patients will be further analysed and divided on the basis of Echocardiography (special scan of the heart that looks at the contraction, relaxation, and the flow of blood in the heart chambers) results into two groups.

1. Those who have impaired contraction (systolic) function of there Left ventricle (left side chamber of the heart)
2. Those who have normal contraction (systolic) function of the left ventricle.

Case notes of these patients will then be studied in detail with regards to their initial presentation, clinical examination, Electrocardiogram (electrical tracing of the heart) and chest X ray (picture of the heart and lungs) report.

These will be co-related with the findings and report of the Echocardiogram.

Once the diagnosis is established, uptake of evidence based medications (beta blockers, ACE inhibitors, spironolactone) and their titration up to the target dose at subsequent follow up visits in the heart failure clinic will be examined.

B) Phase 2 (General practice/ surgery phase)

This part of the study will be conducted at the GP surgery of the identified patient. This will involve accessing the data held at the GP practice with regards to

1. Was heart failure treatment continued after discharge from the hospital clinic?
2. If medications continued then for how long?
3. If medications discontinued then why and by whom (Hospital/GP)?
4. Current medications and the doses
5. Admissions to the hospital if any?
6. Any other co morbidities developed since discharge for the HF clinic?
7. Outcome in terms of mortality
8. The cause of death as specified on the death certificate

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over attending heart failure clinic between 01/01/2002- 31/12/07

Exclusion Criteria:

* less than 18 years.

Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care one stop diagnostic heart failure clinic
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajender Singh, MD, Principal Investigator — county durham and darlington NHS trust
Locations (1):
- Darlington Memorial Hospital, Darlington, Durham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred to the one stop diagnostic heart failure clinic from Jan 2002 to Dec 2007, were followed up till Aug 2011.
Period: Overall Study
Arm/Group | Systolic Dysfunction | Distolic Heart Failure
Started | 270 | 243
Completed | 268 | 241
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Systolic Dysfunction | Distolic Heart Failure | Total
Number analyzed (Participants) | 268 | 241 | 509
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 21 | 70
  >=65 years | 219 | 220 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (10) | 78 (8) | 76 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 157 | 261
  Male | 164 | 84 | 248
Region of Enrollment [Number; unit: participants]
  United Kingdom | 268 | 241 | 509

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Time Frame: Patients would be followed up for average of 7 years
Measure: Number; unit: participants
Arm/Group | Systolic Dysfunction | Distolic Heart Failure
Number analyzed (Participants) | 268 | 241
participants | 163 | 118

2. Secondary Outcome: Cardiovascular Mortality
Time Frame: Patients would be followed up for average of 7years
Measure: Number; unit: participants
Arm/Group | Systolic Dysfunction | Distolic Heart Failure
Number analyzed (Participants) | 268 | 241
participants | 113 [0.315 to 0.610] | 51

3. Secondary Outcome: Admission to Hospital for Any Cause
Description: Number of patients admitted to the hospital will be recorded
Time Frame: During the follow up period of 7 years
Measure: Number; unit: participants
Arm/Group | Systolic Dysfunction | Distolic Heart Failure
Number analyzed (Participants) | 268 | 241
participants | 189 [0.292 to 0.519] | 158 [0.292 to 0.519]

ADVERSE EVENTS:
Arm/Group | Systolic Dysfunction | Distolic Heart Failure
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes